CLINICAL TRIAL: NCT01381874
Title: Randomized, Open-Label Study of Abiraterone Acetate (JNJ-212082) Plus Prednisone With or Without Exemestane in Postmenopausal Women With ER+ Metastatic Breast Cancer Progressing After Letrozole or Anastrozole Therapy
Brief Title: A Study of Abiraterone Acetate Plus Prednisone With or Without Exemestane in Postmenopausal Women With Estrogen Receptor-Positive (ER+) Metastatic Breast Cancer Progressing After Letrozole or Anastrozole Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018286; 212082BCA2001 (Other: Janssen Research & Development, LLC); 2011-000621-80 (EudraCT Number); NCT01355770 (obsolete NCT alias)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Metastatic ER+ Her2- Breast Cancer; Postmenopausal
Keywords: Breast cancer; Abiraterone; Postmenopausal; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — exemestane; Abiraterone Acetate; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Abiraterone acetate + Prednisone or Prednisolone (Experimental): Abiraterone acetate + Prednisone or Prednisolone Abiraterone acetate type=equal unit=mg number=250 form=tablet route=oral use 4 tablets Prednisone or Prednisolone type=equal unit=mg number=5 form=tablet route=oral use. All drugs are taken once daily.
  Interventions: Drug: Abiraterone acetate + Prednisone or Prednisolone
- Abiraterone acetate + Prednisone/Prednisolone + Exemestane (Experimental): Abiraterone acetate + Prednisone/Prednisolone + Exemestane Abiraterone acetate type=equal unit=mg number=250 form=tablet route=oral use 4 tablets Prednisone or Prednisolone type=equal unit=mg number=5 form=tablet route=oral use Exemestane type=equal unit=mg number=25 form=tablet route=oral use. All drugs are taken once daily.
  Interventions: Drug: Abiraterone acetate + Prednisone/ Prednisolone + Exemestane
- Exemestane (Experimental): Exemestane Exemestane type=equal unit=mg number=25 form=tablet route=oral use. All drugs are taken once daily.
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Exemestane — Abiraterone acetate, type=equal, unit=mg, number=250, form=tablet, route=oral use, 4 tablets
  Arms: Exemestane
Drug: Abiraterone acetate + Prednisone/ Prednisolone + Exemestane — Prednisone or Prednisolone, type=equal, unit=mg, number=5, form=tablet, route=oral use. All drugs are taken once daily.
  Arms: Abiraterone acetate + Prednisone/Prednisolone + Exemestane
Drug: Abiraterone acetate + Prednisone or Prednisolone — Abiraterone acetate, type=equal, unit=mg, number=250, form=tablet, route=oral use, 4 tablets
  Arms: Abiraterone acetate + Prednisone or Prednisolone

SUMMARY:
The purpose of this study is to assess the safety and efficacy of oral abiraterone acetate plus oral prednisone and oral abiraterone acetate plus oral prednisone plus oral exemestane, each compared with oral exemestane alone, in postmenopausal women with estrogen receptor-positive (ER+) metastatic (spreading) breast cancer that has relapsed after treatment with letrozole or anastrozole.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (all participants will know the identity of the assigned study drug) study divided into three phases, screening, treatment, and follow-up. During screening, potential patients will be assessed for study eligibility after providing signed informed consent. The treatment phase will comprise a series of 28-day cycles with continuous study treatment until breast cancer progression, when an end-of-treatment visit will be completed before the follow-up phase begins. The duration of participation in the study for an individual patient may be up to approximately 7 years, including follow-up evaluations. Patients will be evaluated for the safety and effectiveness of study treatments. During the treatment phase, patients will take the following study drugs by mouth once daily: abiraterone acetate, 1 g/day, as four 250-mg tablets, on an empty stomach, and patients must not eat for at least 1 hour after abiraterone acetate; prednisone (prednisolone when prednisone is not available), 5 mg/day; and exemestane, 25 mg/day, as a single tablet. The treatment phase will consist of a series of 28-day cycles with continuous study treatment until breast cancer progression. At the planned interim analysis, the Data Review Committee has recommended that further randomization to the abiraterone acetate alone group be stopped and that the study is to be continued otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must be postmenopausal
* ER+, Human epidermal growth factor receptor 2 (Her2) negative metastatic breast cancer
* Disease must have been sensitive to anastrozole or letrozole therapy prior to disease progression
* No more than two prior lines of therapy in the metastatic setting, of which no more than one was chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status score of <=1
* Patients with disease confined only to bone may be included, but patients with purely sclerotic lesions may not participate in the study

Exclusion Criteria:

* Prior treatment with exemestane, ketoconazole, aminoglutethimide, or a CYP17 inhibitor. Prior treatment with ketoconazole for <= 7 days is permitted and topical formulations of ketoconazole are permitted
* Potential patients must not have taken anastrozole, letrozole, fulvestrant, or any chemotherapy for at least 2 weeks (bevacizumab for at least 3 weeks) before randomization
* Anticancer immunotherapy or investigational agent within 4 weeks before randomization, or anticancer radiotherapy (except palliative) or anticancer endocrine therapy within 2 weeks before randomization
* Serious or uncontrolled nonmalignant disease, including active or uncontrolled infection
* Clinical or biochemical evidence of hyperaldosteronism or hypopituitarism
* Any condition that, in the opinion of the investigator, would compromise the well-being of the patient or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (81):
- United States (24):
  - Muscle Shoals, Alabama
  - Fresno, California
  - Los Angeles, California
  - Monterey, California
  - Chicago, Illinois
  - Waterville, Maine
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Henderson, Nevada
  - East Syracuse, New York
  - Johnson City, New York
  - New York, New York
  - Durham, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Portland, Oregon
  - Sioux Falls, South Dakota
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Tyler, Texas
  - Seattle, Washington
- Belgium (9):
  - Antwerp
  - Brussels
  - Duffel
  - Edegem
  - Ghent
  - Hasselt
  - Leuven
  - Liège
  - Wilrijk
- France (5):
  - Bordeaux
  - Caen
  - Pierre-Bénite
  - Saint-Cloud
  - Saint-Herblain
- Ireland (2):
  - Galway
  - Limerick
- Luxembourg (2):
  - Luxembourg
  - Niedercorn
- Netherlands (7):
  - Alkmaar
  - Amsterdam
  - Heerlen
  - Leeuwarden
  - Leiden
  - Rotterdam
  - Sittard
- Poland (2):
  - Bialystok
  - Warsaw
- Russia (8):
  - Chelyabinsk
  - Kazan'
  - Leningrad Region
  - Moscow
  - Saint Petersburg
  - Sochi
  - Stavropol
  - Vladimir
- South Korea (3):
  - Busan
  - Seoul
  - Suwon
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Ukraine (7):
  - Cherkasy
  - Chernivtsi
  - Dnipro
  - Donetsk
  - Kharkiv
  - Odesa
  - Uzhhorod
- United Kingdom (8):
  - Bath
  - Birmingham
  - Exeter
  - London
  - Nottingham
  - Plymouth
  - Sheffield
  - Sutton

REFERENCES:
- [Derived] O'Shaughnessy J, Campone M, Brain E, Neven P, Hayes D, Bondarenko I, Griffin TW, Martin J, De Porre P, Kheoh T, Yu MK, Peng W, Johnston S. Abiraterone acetate, exemestane or the combination in postmenopausal patients with estrogen receptor-positive metastatic breast cancer. Ann Oncol. 2016 Jan;27(1):106-13. doi: 10.1093/annonc/mdv487. Epub 2015 Oct 26. PMID 26504153

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: Participants received exemestane tablet as oral dose of 25 milligram (mg) per day in 28-day treatment cycles until disease progression, unacceptable toxicity, or death (up to 3 years).
- Abiraterone Acetate + Prednisone: Participants received abiraterone acetate tablet at a total oral dose of 1000 milligram (mg) along with 5 mg capsule of prednisone/prednisolone per day in 28-day treatment cycles until disease progression, unacceptable toxicity, or death (up to 3 years).
- Abiraterone Acetate + Exemestane + Prednisone: Participants received abiraterone acetate tablet at a total oral dose of 1000 mg and 5 mg capsule of prednisone/prednisolone along with exemestane tablet 25 mg per day in 28-day treatment cycles until disease progression, unacceptable toxicity, or death (up to 3 years).
Period: Overall Study
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Started | 102 | 89 | 106
Treated | 102 | 87 | 104
Completed | 25 | 26 | 30
Not Completed | 77 | 63 | 76
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 10 | 9
Not completed — Other | 67 | 52 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone | Total
Number analyzed (Participants) | 102 | 89 | 106 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (8.55) | 63.1 (9.17) | 63.8 (10.91) | 62.9 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 89 | 106 | 297
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 84 | 72 | 95 | 251
  Unknown or Not Reported | 18 | 15 | 10 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 92 | 76 | 96 | 264
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 9 | 11 | 4 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 9 | 11 | 8 | 28
  Belgium | 18 | 21 | 21 | 60
  France | 17 | 13 | 11 | 41
  Spain | 11 | 7 | 12 | 30
  United Kingdom | 7 | 12 | 11 | 30
  Italy | 0 | 1 | 4 | 5
  Korea, Republic Of | 1 | 0 | 5 | 6
  Netherlands | 8 | 5 | 8 | 21
  Russia | 20 | 12 | 19 | 51
  Ukraine | 11 | 7 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to first occurrence of disease progression (either radiographic or clinical), or death from any cause. PFS was determined using radiographic progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) on measurable lesions captured by computed tomography (CT) or magnetic resonance imaging (MRI). Clinical disease progression was considered only when disease progression could not be confirmed by CT or MRI, such as when the disease site is skin, bone marrow, or central nervous system.
Time Frame: Approximately 2 years
Population: Intent-to-Treat (ITT) analysis set included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 102 | 89 | 106
Months | 3.68 [1.94 to 5.26] | 3.65 [2.73 to 5.59] | 4.47 [3.68 to 5.59]
Statistical Analysis 1: Comparison: Exemestane vs Abiraterone Acetate + Prednisone; Test type: Superiority; p = 0.437, stratified log-rank test; Hazard Ratio (HR) = 1.143, 95% CI 2-sided [0.816 to 1.603]
Statistical Analysis 2: Comparison: Exemestane vs Abiraterone Acetate + Exemestane + Prednisone; Test type: Superiority; p = 0.794, stratified log-rank test; Hazard Ratio (HR) = 0.958, 95% CI 2-sided [0.695 to 1.320]

2. Primary Outcome: Overall Survival (OS)
Description: OS was calculated as the time from randomization to death from any cause.
Time Frame: Approximately 3 years
Population: ITT analysis set included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 102 | 89 | 106
Months | NA [NA to NA] — Here 'NA' represents that median, lower limit and upper limit of confidence interval (CI) was not estimable due to lesser number of events (high rate of censoring). | 26.41 [23.49 to NA] — Here 'NA' represents that upper limit of CI was not estimable due to lesser number of events (high rate of censoring). | NA [23.79 to NA] — Here 'NA' represents that median and upper limit of CI was not estimable due to lesser number of events (high rate of censoring).
Statistical Analysis 1: Comparison: Exemestane vs Abiraterone Acetate + Prednisone; Test type: Superiority; p = 0.807, stratified log-rank test; Hazard Ratio (HR) = 1.074, 95% CI 2-sided [0.608 to 1.896]
Statistical Analysis 2: Comparison: Exemestane vs Abiraterone Acetate + Exemestane + Prednisone; Test type: Superiority; p = 0.542, stratified log-rank test; Hazard Ratio (HR) = 1.183, 95% CI 2-sided [0.688 to 2.036]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the percentage of participants with measurable disease achieving a best overall response of either complete response (CR) or partial response (PR) based on RECIST. CR: disappearance of all target lesions and non-target lesions. PR: at least a 30 percent (%) decrease in the sum of longest diameter (LD) of target lesions or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Approximately 2 years
Population: ITT analysis set with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 63 | 52 | 66
Percentage of participants | 6.3 | 5.8 | 12.1
Statistical Analysis 1: Comparison: Exemestane vs Abiraterone Acetate + Prednisone; Test type: Superiority; p = 1.000, Fisher Exact; Risk Ratio (RR) = 0.909, 95% CI 2-sided [0.213 to 3.878]
Statistical Analysis 2: Comparison: Exemestane vs Abiraterone Acetate + Exemestane + Prednisone; Test type: Superiority; p = 0.366, Fisher Exact; Risk Ratio (RR) = 1.909, 95% CI 2-sided [0.605 to 6.026]

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of participants with measurable disease achieving a best overall response of a CR, PR, or stable disease (SD) for at least 6 months based on RECIST. Stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study and persistence of one or more non-target lesion(s) and/or maintenance of tumour marker level above the normal limits.
Time Frame: Approximately 2 years
Population: ITT analysis set with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 63 | 52 | 66
Percentage of participants | 12.7 | 9.6 | 22.7
Statistical Analysis 1: Comparison: Exemestane vs Abiraterone Acetate + Prednisone; Test type: Superiority; p = 0.603, Chi-squared; Risk Ratio (RR) = 0.757, 95% CI 2-sided [0.264 to 2.175]
Statistical Analysis 2: Comparison: Exemestane vs Abiraterone Acetate + Exemestane + Prednisone; Test type: Superiority; p = 0.137, Chi-squared; Risk Ratio (RR) = 1.790, 95% CI 2-sided [0.816 to 3.926]

5. Secondary Outcome: Duration of Response
Description: Duration of objective response was measured from the first time that the CR or PR was achieved to the first observation of disease progression (either radiographic or clinical) based on the RECIST criteria.
Time Frame: Approximately 2 years
Population: ITT analysis set with measurable disease at baseline with complete or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 4 | 3 | 8
months | 6.47 [NA to NA] — Here 'NA' represents that lower limit and upper limit of CI was not estimable due to lesser number of events (high rate of censoring). | 4.86 [4.63 to NA] — Here 'NA' represents that upper limit of CI was not estimable due to lesser number of events (high rate of censoring). | 6.93 [4.57 to NA] — Here 'NA' represents that upper limit of CI was not estimable due to lesser number of events (high rate of censoring).

6. Secondary Outcome: Change From Baseline in Serum Endocrine Biomarkers (Estradiol and Estrone) at End of Treatment
Description: Change from baseline in serum endocrine biomarkers (estradiol and estrone) was summarized by treatment at end of treatment.
Time Frame: Baseline and End of treatment (approximately 2 years)
Population: ITT analysis set with valid baseline value and at least 1 post baseline value. Here "n" (number analyzed)" signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: Picomoles Per Liter (Pmol/L)
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 50 | 49 | 56
Picomoles Per Liter (Pmol/L)
  Estradiol | 1.53 (27.643) | -3.35 (13.634) | -1.04 (20.146)
  Estrone: number analyzed (Participants) | 46 | 49 | 56
  Estrone | -34.20 (83.770) | -28.09 (47.779) | -30.60 (42.385)

7. Secondary Outcome: Change From Baseline in Serum Endocrine Biomarkers (Progesterone and Testosterone) at End of Treatment
Description: Change from baseline in serum endocrine biomarkers (Progesterone and Testosterone) was summarized by treatment at end of treatment.
Time Frame: Baseline and End of treatment (approximately 2 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Nanomoles Per Liter (nmol/L)
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
Number analyzed (Participants) | 53 | 50 | 56
Nanomoles Per Liter (nmol/L)
  Progesterone: number analyzed (Participants) | 15 | 8 | 15
  Progesterone | -4.80 (18.268) | 8.98 (15.113) | 12.34 (16.967)
  Testosterone | -0.09 (0.416) | -0.51 (0.459) | -0.48 (0.323)

ADVERSE EVENTS:
Time Frame: Approximately 3 years
Description: Safety population was defined as all randomized participants who received at least one dose of study drug.
Arm/Group | Exemestane | Abiraterone Acetate + Prednisone | Abiraterone Acetate + Exemestane + Prednisone
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/87 | 2/104
Serious Adverse Events (participants affected / at risk) | 12/102 | 18/87 | 28/104
Other Adverse Events (participants affected / at risk) | 79/102 | 76/87 | 84/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=102) | Abiraterone Acetate + Prednisone (N=87) | Abiraterone Acetate + Exemestane + Prednisone (N=104)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoaldosteronism (Endocrine disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 3
Anorectal Varices (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 0 | 1 | 0
Faecal Incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus of Small Bowel (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Asthenia (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 1
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to Peripheral Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to Pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Balance Disorder (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peripheral Artery Stenosis (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=102) | Abiraterone Acetate + Prednisone (N=87) | Abiraterone Acetate + Exemestane + Prednisone (N=104)
Anaemia (Blood and lymphatic system disorders) | 7 | 6 | 9
Abdominal Pain (Gastrointestinal disorders) | 7 | 4 | 14
Constipation (Gastrointestinal disorders) | 9 | 14 | 15
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 13
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 6
Nausea (Gastrointestinal disorders) | 18 | 21 | 22
Vomiting (Gastrointestinal disorders) | 7 | 12 | 19
Asthenia (General disorders) | 12 | 5 | 9
Fatigue (General disorders) | 27 | 24 | 21
Influenza Like Illness (General disorders) | 7 | 0 | 2
Oedema Peripheral (General disorders) | 7 | 6 | 10
Bronchitis (Infections and infestations) | 4 | 7 | 8
Nasopharyngitis (Infections and infestations) | 11 | 5 | 9
Urinary Tract Infection (Infections and infestations) | 0 | 6 | 6
Alanine Aminotransferase Increased (Investigations) | 7 | 5 | 11
Aspartate Aminotransferase Increased (Investigations) | 8 | 5 | 14
Weight Decreased (Investigations) | 4 | 1 | 8
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 13 | 17
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 19 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 8 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 15 | 17
Bone Pain (Musculoskeletal and connective tissue disorders) | 18 | 13 | 13
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 | 7 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 4 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 7 | 10
Dizziness (Nervous system disorders) | 7 | 4 | 8
Dysgeusia (Nervous system disorders) | 2 | 5 | 1
Headache (Nervous system disorders) | 10 | 6 | 15
Insomnia (Psychiatric disorders) | 9 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 14
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 6
Hot Flush (Vascular disorders) | 14 | 14 | 9
Hypertension (Vascular disorders) | 10 | 7 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT01381874/Prot_000.pdf
  • Statistical Analysis Plan (2013-07-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT01381874/SAP_001.pdf